CLINICAL TRIAL: NCT06885736
Title: LEAN Mass Preservation With Resistance Exercise and Protein During Semaglutide and Tirzepatide Therapy (LEAN-PREP Study)
Brief Title: LEAN Mass Preservation With Resistance Exercise and Protein During Semaglutide/Tirzepatide Therapy
Acronym: LEAN-PREP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer (CMO), Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RA HM-2025-01
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: Obesity, research
MeSH Terms: conditions — Obesity | interventions — Resistance Training; Leucine

STUDY DESIGN:
Intervention Model Description: This will be a 6-month 4 arm (control, resistance exercise, protein intake and resistance exercise + protein intake) randomised controlled trial in people with obesity upon initiation of semaglutide/tirzepatide therapy.
Who Masked: Outcomes Assessor
Masking Description: The researcher and the participant will be blinded to the allocation pattern. It is not possible to blind participants to treatment allocation but people making outcome measurements and performing statistical analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Resistance exercise (Experimental): Participants assigned to the resistance exercise group will be asked to perform exercises 3 times a week for the intervention period. The first 3 sessions of the exercise will be performed under the supervision of a qualified exercise specialist to ensure that the participants are happy with the exercises and are performing them appropriately. These will also be group sessions to encourage participants to build social connections to support them during the intervention. A similar group social session will take place at week 4 and then every 4 weeks of the study to overcome any issues with the exercises and to ensure progression to an appropriate intensity.
  Interventions: Behavioral: Resistance exercise
- Protein Intake (Experimental): The aim of this arm of the intervention is to ensure a protein intake of 1.6g/kg/day, as this was the intake level identified as the level after which no further effect was found on muscle mass in the meta-regression from (Morton et al., 2018). For the initial 2 weeks of the study, we will ask participants to consume 2 protein drinks, containing 25g protein (3g leucine), per day - one in the morning and one in the evening. At this stage, we won't know the magnitude of reduction of protein intake following initiation of semaglutide/tirzepatide treatment. After 2 weeks, when the first assessment of dietary intake after beginning semaglutide/tirzepatide treatment occurs, the additional protein will be based on the amount required to ensure 1.6g/kg/day with an aim to spread protein evenly across the day and aim for at least 25g protein (3g leucine) per meal or snack.
  Interventions: Dietary Supplement: Protein Intake
- Resistance exercise + protein intake (Experimental): Participants in this arm will follow the above resistance exercise and protein intake interventions.
  Interventions: Dietary Supplement: Protein Intake; Combination Product: Resistance exercise + protein intake
- Control (No Intervention): Participants assigned to the control group will be asked to maintain their usual exercise habits

INTERVENTIONS:
Behavioral: Resistance exercise — Participants assigned to the resistance exercise group will be asked to perform exercises 3 times a week for the intervention period. The first 3 sessions of the exercise will be performed under the supervision of a qualified exercise specialist to ensure that the participants are happy with the exercises and are performing them appropriately. These will also be group sessions to encourage participants to build social connections to support them during the intervention. A similar group social session will take place at week 4 and then every 4 weeks of the study to overcome any issues with the exercises and to ensure progression to an appropriate intensity.
  Arms: Resistance exercise
Dietary Supplement: Protein Intake — The aim of this arm of the intervention is to ensure a protein intake of 1.6g/kg/day, as this was the intake level identified as the level after which no further effect was found on muscle mass in the meta-regression from (Morton et al., 2018). For the initial 2 weeks of the study, we will ask participants to consume 2 protein drinks, containing 25g protein (3g leucine), per day - one in the morning and one in the evening. At this stage, we won't know the magnitude of reduction of protein intake following initiation of semaglutide/tirzepatide treatment. After 2 weeks, when the first assessment of dietary intake after beginning semaglutide/tirzepatide treatment occurs, the additional protein will be based on the amount required to ensure 1.6g/kg/day with an aim to spread protein evenly across the day and aim for at least 25g protein (3g leucine) per meal or snack.
  Other Names: leucine
  Arms: Protein Intake; Resistance exercise + protein intake
Combination Product: Resistance exercise + protein intake — Participants in this arm will follow the above resistance exercise and protein intake interventions
  Arms: Resistance exercise + protein intake

SUMMARY:
The aim of the current study is to determine whether resistance exercise and/or protein intake can preserve lean mass and improve physical function in patients with obesity initiating semaglutide/tirzepatide therapy. To achieve this aim the study will have the following objectives.

In people with obesity initiating semaglutide/tirzepatide therapy

1. Form a PPI group to refine the study protocol and establish study materials,
2. Quantify the effects of a pragmatic resistance exercise intervention and/or increasing protein intake on lean mass and physical function during semaglutide/tirzepatide induced weight loss,
3. Establish whether the resistance exercise intervention and/or increasing protein intake has concomitant benefits on glycaemic control, lipids, liver function, quality of life, physical activity and sleep during semaglutide/tirzepatide induced weight loss.

The participants will:

Begin their weight loss medication, starting at a low dose and then increasing the dose to maximize weight loss. They will be randomly assigned by a computer to ONE of the following groups and will be followed up to 6-months:

* Control group
* Protein intake group
* Muscle strengthening exercise group
* Muscle strengthening exercise AND protein intake group.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* BMI 27-45

Exclusion Criteria:

* Currently or in the past 6 months participating in any vigorous aerobic activity (>1h per week) or any resistance exercise.
* BP of 160/100mmHg or higher
* Insulin therapy
* Any known medical condition that prevents participants from exercising safely
* A personal or family history of medullary thyroid carcinoma
* Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* History of chronic or acute pancreatitis
* History of proliferative diabetic retinopathy or diabetic maculopathy
* History of ketoacidosis or hyperosmolar state/coma
* History of severe hypoglycaemia and/or hypoglycaemia unawareness within last 6 onths
* Clinically significant gastric emptying abnormality or have undergone or plan to undergo gastric bypass or restrictive bariatric surgery or chronically taking drugs that directly affect GI motility
* Any of the following CV conditions in last 2 months: acute MI, stroke or hospitilisation due to CHF
* History of NYHA IV CHF
* Acute or chronic hepatitits, signs and symptoms of any liver disease other than NAFLD, ALT > 3 times the upper limit of normal
* eGFR <45mL/min/1.73m2
* Significant uncontrolled endocrine abnormaility in the opinion of clinical investigator
* Serum calcitonin >35ng/L
* Evidence of active autoimmune abnormality that is likely to requite systemic glucocorticoid treatment in the next 12 months
* Had or waiting for an organ transplant
* History of an active or untreated malignancy or in remission from a clinically significant malignancy for less than 5 years
* Any other aspect of history or condition that may limit the ability of the patient to complete the study
* Having been treated with prescription drugs that promote weight loss in the last 3 months
* Receiving chronic systemic glucocorticoid therapy within last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI measured quadriceps cross sectional area (CSA) | From enrollment (at baseline) to the end of treatment at 6 months.
  At the mid-point of the thigh, we will measure the cross-sectional area of the quadriceps muscle and quantify muscle's thickness and size.

SECONDARY OUTCOMES:
MRI measured liver fat | From enrollment (at baseline) to the end of treatment at 6 months.
  We will also assess liver fat using an IDEAL scan.
MRI measured intramuscular fat content (total thigh) | From enrollment (at baseline) to the end of treatment at 6 months.
  We will quantify intramuscular fat content
Muscle strength | From enrollment (at baseline) to the end of treatment at 6 months.
  Grip strength will be measured 3 times in each hand using a Jamar dynamometer.
Energy intake | From enrollment (at baseline) to the end of treatment at 6 months.
  Baseline energy intake will be quantified by the use of the EPIC food frequency questionnaire and multi-pass 24h recall. Further 24h recalls will be carried out at 0.5,1,3 and 6 months of the follow up period.
Physical activity and sleep levels | From enrollment (at baseline) to the end of treatment at 6 months.
  Participants will be asked to wear and accelerometer for a 7-day period to quantify physical activity and sedentary behaviour. The accelerometer is a wrist born watch and we will ask participants to wear this device for 24h a day for the 7-day measurement period. We will use tri-axial accelerometers and following data collection we will process the accelerometer counts using R software and generate the daily amount of light, moderate and vigorous physical activity along with sleep.
Activities of Daily Living | From enrollment (at baseline) to the end of treatment at 6 months.
  This will be quantified by the Barthel activities of daily living questionnaire.
Whole blood glycated haemoglobin (HbA1c) | From enrollment (at baseline) to the end of treatment at 6 months.
Oral glucose tolerance test | From enrollment (at baseline) to the end of treatment at 6 months.
  An oral glucose tolerance test will be performed with a cannula inserted and a baseline blood sample collected, a 75g glucose load consumed and further samples collected at 15, 30, 60 90 and 120 min. Samples will be analysed for glucose and insulin levels.
Blood lipids | From enrollment (at baseline) to the end of treatment at 6 months.
Liver function | From enrollment (at baseline) to the end of treatment at 6 months.
  We will measure aspartate amino transferase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), albumin (ALB), total protein (TP), gamma-glutamyltransferase (GGT) and bilirubin.
Plasma GLP-1 and GIP | From enrollment (at baseline) to the end of treatment at 6 months.
Concomitant medication | From enrollment (at baseline) to the end of treatment at 6 months.
Fib-4 score | From enrollment (at baseline) to the end of treatment at 6 months.
  Fib-4 score will be calculated from liver function test
hsCRP | From enrollment (at baseline) to the end of treatment at 6 months.
IL-6, IL-10, IL1Ra and TNF-alpha. | From enrollment (at baseline) to the end of treatment at 6 months.
Gait Speed | From enrollment (at baseline) to the end of treatment at 6 months.
  Habitual gait speed will be measured during a 4 metre walk test
Chair rise performance | From enrollment (at baseline) to the end of treatment at 6 months.
  The number of chair rises completed in 30 seconds measured.
Aerobic Fitness | From enrollment (at baseline) to the end of treatment at 6 months.
  Aerobic fitness will be quantified with the 6 min walk test.
Macronutrient Intake | From enrollment (at baseline) to the end of treatment at 6 months.
  Baseline carbodhyrate, fat and protein intake (all g/day) will be quantified by the use of the EPIC food frequency questionnaire and multi-pass 24h recall. Further 24h recalls will be carried out at 0.5,1,3 and 6 months of the follow up period.
Quality of Life assessed using the EQ-5D-5L questionnaire | From enrollment (at baseline) to the end of treatment at 6 months.
  This will be quantified by the EQ-5D-5L questionnaire.
Body Composition via DEXA scan | From enrollment (at baseline) to the end of treatment at 6 months.
  fat and fat free mass via Dual Energy X-ray Absorptiometry (DEXA)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morton RW, Murphy KT, McKellar SR, Schoenfeld BJ, Henselmans M, Helms E, Aragon AA, Devries MC, Banfield L, Krieger JW, Phillips SM. A systematic review, meta-analysis and meta-regression of the effect of protein supplementation on resistance training-induced gains in muscle mass and strength in healthy adults. Br J Sports Med. 2018 Mar;52(6):376-384. doi: 10.1136/bjsports-2017-097608. Epub 2017 Jul 11. PMID 28698222
- [Background] Mettler S, Mitchell N, Tipton KD. Increased protein intake reduces lean body mass loss during weight loss in athletes. Med Sci Sports Exerc. 2010 Feb;42(2):326-37. doi: 10.1249/MSS.0b013e3181b2ef8e. PMID 19927027
- [Background] Lundgren JR, Janus C, Jensen SBK, Juhl CR, Olsen LM, Christensen RM, Svane MS, Bandholm T, Bojsen-Moller KN, Blond MB, Jensen JB, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Healthy Weight Loss Maintenance with Exercise, Liraglutide, or Both Combined. N Engl J Med. 2021 May 6;384(18):1719-1730. doi: 10.1056/NEJMoa2028198. PMID 33951361
- [Background] Westcott WL. Resistance training is medicine: effects of strength training on health. Curr Sports Med Rep. 2012 Jul-Aug;11(4):209-16. doi: 10.1249/JSR.0b013e31825dabb8. PMID 22777332
- [Background] Umpierre D, Ribeiro PA, Kramer CK, Leitao CB, Zucatti AT, Azevedo MJ, Gross JL, Ribeiro JP, Schaan BD. Physical activity advice only or structured exercise training and association with HbA1c levels in type 2 diabetes: a systematic review and meta-analysis. JAMA. 2011 May 4;305(17):1790-9. doi: 10.1001/jama.2011.576. PMID 21540423
- [Background] Al Ozairi E, Alsaeed D, Al Roudhan D, Jalali M, Mashankar A, Taliping D, Abdulla A, Gill JMR, Sattar N, Welsh P, Gray SR. The effect of home-based resistance exercise training in people with type 2 diabetes: A randomized controlled trial. Diabetes Metab Res Rev. 2023 Oct;39(7):e3677. doi: 10.1002/dmrr.3677. Epub 2023 Jun 17. PMID 37330638
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28698222/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19927027/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33951361/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22777332/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21540423/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37330638/